CLINICAL TRIAL: NCT07398131
Title: Voice-Induced Motor Intention to Enhance Upper Limb Rehabilitation Efficacy of Exoskeleton Robots for Stroke Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Hospital, Ministry of Health and Welfare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TYGH114109
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: To Understand Whether Increasing the Willingness to Exercise Can Improve Rehabilitation Outcomes (Upper Limb Motor Activation); for Patient With Stroke
Keywords: upper limb motor activation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Voice-Enhanced Motor Imagery Group (Experimental): Participants in this group receive upper limb rehabilitation using the Nimbo single-joint robot combined with an "Active Imagery" protocol. Before each movement, patients focus on imagining the target action for 2 seconds and then issue a standardized voice command (e.g., "bend hand") to trigger the robotic assistance. The training is conducted for 30 minutes per session, 5 sessions per week, for a total of 4 weeks.
  Interventions: Device: single-joint robot (Passive Mode)
- Passive Robotic Training Group (Active Comparator): Participants in this group receive conventional passive robotic-assisted rehabilitation using the Nimbo single-joint robot. The robot moves the patient's limb through a preset range of motion automatically. There is no requirement for synchronized motor imagery or voice commands during the session. The training frequency and duration are identical to the experimental group: 30 minutes per session, 5 sessions per week, for 4 weeks.
  Interventions: Device: single-joint robot (Active Voice-Controlled Mode)

INTERVENTIONS:
Device: single-joint robot (Active Voice-Controlled Mode) — A robotic exoskeleton used with a voice-trigger interface. Patients perform motor imagery for 2 seconds followed by a voice command to activate the device.
  Arms: Passive Robotic Training Group
Device: single-joint robot (Passive Mode) — The same robotic exoskeleton used in a traditional passive rehabilitation mode where the device moves the limb automatically according to preset parameters.
  Arms: Voice-Enhanced Motor Imagery Group

SUMMARY:
This study aims to investigate whether combining "motor imagery" (the mental visualization of movement) with robotic exoskeleton therapy can improve upper limb recovery in stroke patients. Conventional robotic therapy often involves passive movement driven by the machine. In this study, patients in the experimental group will use their own voice to trigger the robot (e.g., saying "bend arm") while simultaneously imagining the movement. The research will compare this voice-enhanced "active" approach with traditional passive robotic training to see if it better promotes brain-to-muscle signal recovery and improves overall arm function .

DETAILED DESCRIPTION:
Background and Rationale: Stroke is a leading cause of adult disability, and the "golden period" for rehabilitation requires intensive therapy to trigger muscle movement. Recent theories suggest that combining motor imagery with physical activity-known as Brain-Computer Interface (BCI) concepts-may be more effective than passive movement alone. However, complex EEG-based BCI is difficult to implement clinically. This study proposes a simplified "voice-controlled" interface to simulate the motor intent-to-action loop.

Study Design: This is a randomized, assessor-blinded, parallel-group clinical trial involving 32 subacute or chronic stroke patients. Participants will be randomly assigned to one of two groups for a 4-week intervention (5 sessions per week, 30 minutes per session).

Interventions:

Experimental Group (Voice + Exoskeleton): Patients will use the Nimbo single-joint robot. Before each movement, they will focus on imagining the target action for 2 seconds, then issue a standardized voice command (e.g., "bend hand") to trigger the robotic assistance.

Control Group (Passive Exoskeleton): Patients will receive conventional robotic-assisted training where the Nimbo exoskeleton moves the limb through a preset path without voice prompts or intentional imagery requirements.

Outcome Measures: Evaluations will be conducted at baseline (T0), week 2 (T1), and week 4 (T2).

Primary Outcome: Upper limb motor function measured by the Fugl-Meyer Assessment - Upper Extremity (FMA-UE).

Secondary Outcomes: Brunnstrom stage (recovery phase), KVIQ-10 (subjective imagery), Laterality Judgment Task (objective imagery processing), Sense of Agency (SoA) questionnaire, and System Usability Scale (SUS).

Safety and Monitoring: Safety checks, including pain (NRS), fatigue (RPE), and skin inspections, will be performed after every session. Any adverse events will be reported to the Institutional Review Board (IRB) and data safety monitoring personnel .

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke diagnosed by CT or MRI
* Stroke onset occurred at least 1 month prior to enrollment
* Aged 20 to 80 years
* Moderate to severe upper limb impairment (Fugl-Meyer Assessment-Upper Extremity score between 13 and 47)
* Cognitive function sufficient to follow instructions (MMSE score > 20)
* Stable medical condition with no severe pain in the affected upper limb

Exclusion Criteria:

* Severe spasticity of the affected upper limb (Modified Ashworth Scale score > 2)
* History of other neurological diseases (e.g., Parkinson's disease, brain tumor)
* Serious orthopedic conditions or skin lesions on the affected upper limb that prevent robot use
* Unstable epilepsy or severe psychiatric disorders
* Pregnancy

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment - Upper Extremity (FMA-UE) | Baseline (T0), 2 weeks (T1), and 4 weeks (T2).
  A quantitative measure of upper limb motor recovery. The scale includes 33 items assessing reflexes, movement patterns, and coordination. Scores range from 0 to 66, with higher scores indicating better motor function.

SECONDARY OUTCOMES:
Brunnstrom Recovery Stage (Upper Limb) | Baseline (T0), 2 weeks (T1), and 4 weeks (T2).
  A 6-stage classification system used to categorize the degree of motor recovery in post-stroke hemiplegia, ranging from Stage I (flaccidity) to Stage VI (normal motor function).
Kinesthetic and Visual Imagery Questionnaire (KVIQ-10) | Baseline (T0), 2 weeks (T1), and 4 weeks (T2).
  Evaluates the clarity of visual imagery and intensity of kinesthetic imagery on a 5-point scale. Scores range from 10 to 50; higher scores indicate better imagery ability.
Laterality Judgment Task (LJT) - Accuracy and Reaction Time | Baseline (T0), 2 weeks (T1), and 4 weeks (T2).
  Measures the mental rotation ability by identifying the laterality (left/right) of hand images. Accuracy (percentage) and reaction time (seconds) are recorded.
Sense of Agency (SoA) Questionnaire | Baseline (T0), 2 weeks (T1), and 4 weeks (T2).
  This questionnaire assesses the patient's subjective feeling of control over the robotic movement. It consists of 4 items scored on a 7-point Likert scale, ranging from -3 (strongly disagree) to +3 (strongly agree). The total score is the sum of all items, ranging from -12 to +12. Higher scores indicate a stronger sense of agency (a greater feeling of being the cause of the robotic movement).
System Usability Scale (SUS) | 4 weeks (T2).
  The System Usability Scale (SUS) is a 10-item instrument for evaluating the usability of the voice-controlled robotic interface. Each item is scored on a 5-point scale from 0 (strongly disagree) to 4 (strongly agree). The final score is calculated by multiplying the sum of the item scores by 2.5, resulting in a total score ranging from 0 to 100. Higher scores indicate better usability and higher user satisfaction.